CLINICAL TRIAL: NCT02528448
Title: The Effect of 0,9% NaCl on the Kidney Function, Vasoactive Hormones, Biomarkers and Glycosaminglycanes in Plasma in Patients Operated on for Primary Hiparthrosis
Brief Title: 0,9% NaCl Effect on Kidney Function and Glycocalyx in Patients Operated on for Primary Hiparthrosis
Acronym: KIPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, MD, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NPE-01-2014
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Nephrotoxicity
Keywords: Vasoactive hormones; bio markers; salt regulation; Renal variables
MeSH Terms: interventions — Plasma-lyte 148; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plasma-lyte (Active Comparator): Continuous 1 hour infusion of plasma-lyte 15 micrograms/kg/hour for the first hour then 5 micrograms/kg/hour + amount needet for blood replacement
  Interventions: Drug: Plasma-lyte
- 0,9% saline (Active Comparator): Continuous 1 hour infusion of 0,9% saline15 micrograms/kg/hour for the first hour then 5 micrograms/kg/hour + amount needet for blood replacement
  Interventions: Drug: 0,9% saline

INTERVENTIONS:
Drug: Plasma-lyte — Continuous 1 hour infusion of plasma-lyte 15 micrograms/kg/hour for the first hour then 5 micrograms/kg/hour + amount needet for blood replacement
  Other Names: ATC: B 05 BB 01
  Arms: plasma-lyte
Drug: 0,9% saline — Continuous 1 hour infusion of 0,9% saline 15 micrograms/kg/hour for the first hour then 5 micrograms/kg/hour + amount needet for blood replacement
  Other Names: sodium chloride
  Arms: 0,9% saline

SUMMARY:
The purpose of this study is to determine if chloride is nephrotoxic using 0,9% saline versus Plasma-Lytein in patients having primary hip replacement surgery. The outcome is found measuring bio markers, vasoactive hormones and salt regulation. And to measure syndecan as a marker for glycocalyx degradation.

DETAILED DESCRIPTION:
Hypothesis:

Chloride has a nephrotoxic effect, which can be shown partially by measuring bio markers for tubular injury in urine, partially by the changes in tubular transport of sodium and water in different parts of the nephron. This can be demonstrated using isotone sodium solutions with a lower chloride concentration in this study plasma-lyte versus normal isotone saline.

Klorid has a toxic effect on the glycocalyx layer and leads to a rise in syndecan 1 and simultaneously a change in Salt Blood Test either by a direct simulation and ANP levels in plasma or as a consequence of the hyperchloremic acidosis. This can be demonstrated using isotone sodium solutions with a lower chloride concentration in this study plasma-lyte versus normal isotone saline.

Purpose:

The purpose is to observe changes in bio markers, vasoactive hormones and salt regulation in patients randomized to either 0,9% saline or plasma-lyte undergoing primary uncemented hip replacement surgery.

Design:

40 patients undergoing primary uncemented hip replacement surgery will be randomized to either 0,9% saline or plasma-lyte for standard fluid resuscitation and blood loss replacement in this controlled and double blinded study. The patients will deliver a 24 hour urine sample before surgery and approximately 10 days after. From the start of the surgery and to the day after all urine will be collected and blood samples will be taken.

Perspective:

If chloride is found to be nephrotoxic it could lead to a general change in fluid resuscitation recommendations in critically ill patient, patients with kidney disease and patients undergoing surgery. It will also expand our knowledge about the permeability of the blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Indication for uncemented primary hiparthroplasty
* age < 60

Exclusion Criteria:

* Blooddonation or transfusion during the last month
* Not willing to participate
* estimated GFR below 30ml/min
* type 1 diabetes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Urinary excretion of Neutrophil gelatinase-associated lipocalin | two days

SECONDARY OUTCOMES:
plasma Syndecan-1 | two days
plasma renin concentration | two days
Urinary excretion of cyclic guanosine monophosphate | two days
Urinary excretion of epithelial sodium channels | two days
Urinary excretion of water channels | two days
Plasma concentration of angiotensin 2 | two days
Plasma concentration of aldosterone | two days
Plasma concentration of atrial natriuretic peptide (ANP) | two days
Plasma concentration of brain natriuretic peptide (BNP) | two days
Plasma concentration of cyclic guanosine monophosphate (cGMP) | two days
Plasma concentration of endothelin | two days
Plasma concentration of vasopressin (AVP, ADH) | two days
Urinary excretion of Fatty acid-binding protein | two days
Urinary excretion of Kidney Injury Molecule | two days
Free water clearance | two days
Plasma concentration of albumin | two days
Plasma concentration of chloride | two days
Plasma concentration of creatinine | two days
Plasma osmolarity | two days
Plasma concentration of sodium | two days
Plasma concentration of potassium | two days
Urinary excretion of creatinine | two days
Urinary excretion of chloride | two days
Urinary excretion of sodium | two days
Urinary excretion of potassium | two days
Fractional urinary sodium excretion | two days
Urinary osmolarity | two days
Urinary excretion of albumin | two days
Urinary excretion of sodium-chloride symporter | two days
pH | two days
pulse | two days
middle arterial pressure | two days

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, PhD, Principal Investigator — Regional Hospital Holstebro; Erling B Perdersen, MD, DMSc, Study Director — Regional Hospital Holstebro; Niels Peter Ekeløf, MD, PhD, Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Department of Medical Research, Regional Hospital Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Ostergaard AM, Jorgensen AN, Bovling S, Ekelof NP, Mose FH, Bech JN. Effect of 0.9% NaCl compared to plasma-lyte on biomarkers of kidney injury, sodium excretion and tubular transport proteins in patients undergoing primary uncemented hip replacement - a randomized trial. BMC Nephrol. 2021 Mar 26;22(1):111. doi: 10.1186/s12882-021-02310-4. PMID 33771116